CLINICAL TRIAL: NCT07002697
Title: High-Risk Plaques Identification Using Coronary Computed Tomography and Computational Fluid Dynamics
Brief Title: Geometrical Influences on Atherosclerosis and Blood Flow
Status: Recruiting | Type: Observational
Sponsor: Bangladesh University of Engineering and Technology (Other)
Collaborators: National Institute of Cardiovascular Diseases, Bangladesh (Other)
Responsible Party: Principal Investigator, Muhammad Tarik Arafat, Professor, Bangladesh University of Engineering and Technology
Other Study IDs: BUET/ERC/2024/04
Record Dates: First submitted 2025-04-19; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Atherosclerosis and Blood Flow in Coronary Artery
Keywords: Computational Fluid Dynamics (CFD); Design Of Experiment (DOE); Computed Tomography (CT); Acute Coronary Syndrome (ACS)
MeSH Terms: conditions — Atherosclerosis; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who have Acute Coronary Syndrome and did a CT angiogram: In observational studies aimed at identifying high-risk plaques using coronary computed tomography (CT) and computational fluid dynamics (CFD), the group or cohort typically consists of people having diagnostic imaging for suspected or established coronary artery disease (CAD). Participants are frequently chosen based on clinical indicators such as chest discomfort, a history of myocardial infarction, or abnormal stress test findings. Cohort characteristics include age, gender, cardiovascular risk factors (such as hypertension, diabetes, hyperlipidaemia, and smoking), and previous CAD therapies. The study will examine plaque features (e.g., low-attenuation plaques, positive remodelling) and hemodynamic parameters generated from CFD (e.g., wall shear stress, pressure gradients) to stratify risk. Detailed demographic, clinical, and imaging data are collected to examine relationships between plaque features and cardiovascular outcomes, ensuring a thorough analysis.

SUMMARY:
The study investigates the use of advanced imaging techniques and computational methods to identify high-risk plaques in coronary arteries. These plaques are significant because they have the potential to cause acute coronary syndrome (ACS), a condition that includes heart attacks and unstable angina. The research focuses on integrating Coronary Computed Tomography (CCT) with Computational Fluid Dynamics (CFD) to provide detailed insights into plaque characteristics and their hemodynamic environment.

The study's primary aim is to enhance the early detection and characterization of high-risk coronary plaques that could lead to ACS. By combining CCT, a non-invasive imaging technique, with CFD, which stimulates blood flow dynamics, the study seeks to: Identify High-Risk Plaques, Apply CFD to analyze the blood flow around these plaques, Improve Prediction of ACS, Inform Clinical Decision-Making.

Computational fluid dynamics (CFD) analysis of CCT data can also provide a non-invasive hemodynamic assessment to identify high-risk plaques destined to cause acute coronary syndrome. Patients with adverse plaque characteristics like positive remodeling or low-attenuation plaque have a greater risk of future coronary events.

DETAILED DESCRIPTION:
The locally adapted workflow for the identification of high-risk atherosclerotic plaques that may cause Acute Coronary Syndrome (ACS) based on the integration of CCT and CFD is carried out systematically. These are the steps in the presented methodology, namely, the patient cohort, imaging, data handling and analysis, CFD simulation, and clinical implementation.

Firstly, select patients based on symptoms of coronary artery disease (CAD), high-risk factors (e.g., family history, hypertension, diabetes), or those requiring further evaluation after preliminary tests and then Preparation: Give drugs to achieve a proper rate of heartbeat. The order includes checking the patient's habits for proper hydration and contraindications to the use of contrast media. If investigators read this, then follow CCT imaging protocol. Conduct CCT with the help of a multi-detector CT scanner only. Take detailed images of the coronary arteries. Plan to administer iodinated contrast material to improve the visual display of coronary arteries. Moreover, electrocardiographic gating ensures the timely exposure of the patient's heart to radiation during the cardiac cycle to minimize motion. All the above processes have to be accomplished then the remaining work is taken care of by Mimics and Ansys Simulation software. Create reconstructions of the coronary arteries using Ansys software and out of the CCT data that was acquired. Grasp positive remodeling, low attenuation plaque, napkin ring sign, and spotty calcification in atherosclerotic plaques. Document the features that were noticed about the plaques that are in the identified places; the sizes and the shapes and the location certainly. The working process is, to a large extent, sequential. When one of them is absent the other does not work, or does not operate within the protocol, we do not discover our result. Following that, ''Cut out' the coronary artery regions of interest from the reconstructed 3D images. Develop a mesh based on the segmented coronary artery regions. This entails the segmentation of the artery into small parts that are useful in making a CFD analysis. CFD Simulation has some conditions that are important for the results of the research.

Boundary Conditions: Define physiological boundary conditions, such as blood flow rates, pressure, and velocity, based on patient-specific data.

Simulation: Configure the CFD software with the segmented geometry and boundary conditions. Run the CFD simulations to calculate hemodynamic parameters, including wall shear stress (WSS), and flow velocity profiles.

Data Analysis: Analyze the CFD results to understand the hemodynamic environment within the coronary arteries and identify regions with abnormal hemodynamic forces.

After Completing the above processes, Integrate anatomical data from CCT (plaque characteristics) with hemodynamic data from CFD (WSS). Identify high-risk plaques based on combined criteria, including anatomical vulnerability and hemodynamic stress. Then, the investigators Generate a detailed report summarizing the findings from CCT and CFD analysis. The investigators Stratify patients into different risk categories (low, moderate, high) based on the comprehensive assessment. Finally, the investigators will adjust the treatment plan based on the findings and analysis of the patient's response.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-70 years.
* Presenting with symptoms of CAD (e.g., chest pain, shortness of breath) or having multiple risk factors (e.g., hypertension, diabetes, smoking).
* Able to provide informed consent.

Exclusion Criteria:

* Severe renal impairment (due to contrast media risk).
* Previous allergic reaction to iodinated contrast media.
* Pregnant or lactating women.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes patients diagnosed with atherosclerosis, identified through CT angiography (CTA). High-resolution CT scan data reconstruct patient-specific vascular geometries, focusing on regions of clinical interest, such as arterial bifurcations and stenotic segments. Key parameters include Curvature, Surface Roughness, stenosis severity and bifurcation angles, allowing for a detailed computational fluid dynamics (CFD) analysis of hemodynamic forces contributing to endothelial dysfunction and plaque progression.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Geometrical Influences on Atherosclerosis and Blood Flow: A Computational Fluid Dynamics and Experimental Design Approach | Each patient is monitored for upto 1 year after enrollment to assess plaque changes and hemodynamics via periodic imaging and analysis.
  The primary outcome of this study is the focus on evaluating the impact of vascular geometry on blood flow patterns and their role in the development of atherosclerosis. Using Computational Fluid Dynamics (CFD) simulations, the study investigates critical hemodynamic factors, such as wall shear stress, pressure gradients, and recirculation zones, which are influenced by variations in vessel geometry. By integrating experimental data with computational models, the study aims to identify specific geometrical features that contribute to plaque formation and progression, ultimately enhancing the understanding of atherosclerosis and guiding targeted interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tarik Arafat, PhD, Principal Investigator — Department of Biomedical Engineering, Bangladesh University of Engineering and Technology (BUET), Dhaka - 1205; Dr. M G Azam, MBBS, MD, FSCAI, Principal Investigator — NICVD, Dhaka
Locations (1):
- National Institute of Cardiovascular Disease (NICVD), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT07002697/Prot_ICF_000.pdf